CLINICAL TRIAL: NCT02255903
Title: Middle Cerebral To Umbilical Artery Doppler Ratio And Amniotic Fluid Volume Measurement In Post-date Pregnancies in King Faisal Military Central City
Brief Title: Middle Cerebral To Umbilical Artery Doppler Ratio And Amniotic Fluid Volume Measurement In Post-date Pregnancies in King Khalid Military Central City
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, khalid abd aziz mohamed, lecturer and consultant of oblgyne, Benha University
Other Study IDs: khalid-mohamed
Record Dates: First submitted 2014-09-26; First posted 2014-10-03 (Estimated); Last update posted 2022-02-14 (Actual); Status verified 2022-01

CONDITIONS: Pregnancy, Prolonged
MeSH Terms: conditions — Pregnancy, Prolonged | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 1(Control Group):: ultrasound and Doppler examination: of 100 pregnant females with gestational age 37-40 weeks.
  Interventions: Other: ultrasound and Doppler examination
- Group 2 (post date Group): ultrasound and Doppler examination:will be done for 100 pregnant females with gestational age 41 weeks or more
  Interventions: Other: ultrasound and Doppler examination

INTERVENTIONS:
Other: ultrasound and Doppler examination — ultrasound and Doppler examination: Trans-abdominal ultrasound examination will be peformed to all patienst while women in a slightly tilted position with the head of the bed raised 30 degrees and with a small pillow under the right lion

SUMMARY:
The aim of this study is to assess the values of MCA PI / UA PI and MCA RI / UA RI ratios and amniotic fluid volume in predicting the adverse perinatal fetal outcome in uncomplicated postdate pregnancy

DETAILED DESCRIPTION:
The Study Will be a case-control study that will be conducted at Banha University Hospital and AFHSR in Saudi Arabia after the approval of Institutional ethical committee. One hundred pregnant women will be recruited from antenatal clinic. Starting from November 2022. An informed consent will be obtained from the patients . The patients will be subdivided into two groups:

Group 1(Control Group):consist of 100 pregnant females with gestational age 37-40 weeks.

Group 2 (post date Group):consist of 100 pregnant females with gestational age 41 weeks or more.

Inclusion criteria:

1. Singleton, viable fetus in the vertex presentation.
2. History of regular menstrual cycles.
3. Gestational age calculated from the first day of last menstryal period or by first-trimester or second-trimester (before 20 weeks) ultrasound examination.
4. No obstetric or medical complications of pregnancy apart from post-date pregnancy

All patients will be subjected to:

1. Detailed history: including, personal history, menstural history, obstetric history, present history and past history.
2. Physical examination: general, abdominal and pelvic examination.
3. Investigations: including, A- Ultrasound examintion for amniotic fluid index (AFI) measurement.

B- Doppler studies:

i - Middle cerebral artery pulsatility index (MCA -PI) and resistace index(MCA-RI).

ii - Umbilical artery pulsatility index (UA-PI) and resistance index (UA-RI). iii - Cerebro-Placental ratio (CPR).

ELIGIBILITY:
Inclusion Criteria:

1. Singleton, viable fetus in the vertex presentation
2. History of regular menstrual cycles
3. Gestational age calculated from the first day of last menstryal period or by first-trimester or second-trimester (before 20 weeks) ultrasound examination
4. No obstetric or medical complications of pregnancy apart from post-date pregnancy

Exclusion Criteria:

1. Patients unsure of their dates
2. Medical disorders with pregnancy as (hypertension, diabetes mellitus or Rh isoimmunization)
3. Prelabor rupture of membranes
4. Polyhydramnios
5. Women with multiple pregnancy
6. Congenital fetal anomalies
7. Antepartum hemorrhage
8. Previus cesarean section
9. Fetal malpresentation

Ages: 19 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Two hundred pregnant women will be recruited from outpatient clinic. Starting from February 2022. An informed consent will be obtained from the patients . The patients will be subdivided into two groups:
  Group 1(Control Group):consist of 100 pregnant females with gestational age 37-40 weeks.
  Group 2 (post date Group):consist of 100 pregnant females with gestational age 41 weeks or more.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-02 (Estimated); Primary Completion 2023-05 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Adverse pregnancy outcome | at time of delivery

CONTACTS AND LOCATIONS:
Overall Officials: khalid ibrahim, MD, Study Chair — Armed Forces Hospitals, Southern Region, Saudi Arabia; KHALID IBRAHIM, MD, Study Director — Armed Forces Hospitals, Southern Region, Saudi Arabia
Locations (1):
- AFHSR, Khamis Mushait, Afhsa, Saudi Arabia